CLINICAL TRIAL: NCT00232778
Title: A Multicenter Trial of Localized Radiation Therapy to Inhibit Restenosis (GAMMA V)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00-5501
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: GAMMA-Iridium-192 catheter

SUMMARY:
The objectives of this study are:

1. To show a reduction in the late thrombosis (LT) rate following percutaneous revascularization using current interventional techniques with new stent placement and intravascular radiation therapy (IRT) with a long-term antiplatelet regimen (12 months) compared to the stented patients on short-term antiplatelet regimen (2 months) from the IRT arm of GAMMA I Trial.
2. To show equivalence in the LT rate following percutaneous revascularization using current interventional techniques without new stent placement and IRT with a long-term antiplatelet regimen (6 months) compared to non-stented patients on short term antiplatelet therapy (2 months or less) from a pooling of the IRT arms of the GAMMA I, SCRIPPS, and WRIST Trials.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a restenosis of >60% (by subjective angiographic determination of the minimal luminal diameter compared to the distal reference diameter) within a native coronary artery which has previously undergone stent placement.
2. The patient has a history, signs of, or laboratory studies that suggest coronary ischemia attributable to the target stenosis.
3. The study target lesion must be located in a restenotic native coronary artery measuring >2.75 and <4.0 mm in diameter and 45 mm in length. The target lesion must have undergone coronary interventional treatment >4 weeks previously.
4. The vessel 1 cm distal to the target lesion is >2.5 mm in diameter.

5 Patients age must be >18 years and <85 years.

Exclusion Criteria:

1. Attempts to treat lesions in other vessels during the procedure were unsuccessful.
2. The patient sustained a recent (<72 hours) myocardial infarction defined as a serum CK 2x the upper limit of normal and elevated MB.
3. Serum creatinine >2.0 mg/dl.
4. The left ventricular ejection fraction is <40%.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579
Dates: Start 2000-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness parameters will be late thrombosis of the target lesion at
9 months for non-stented patients and late thrombosis of the target lesion at
15 months for stented patients.
The safety criteria will include post-procedure Q-wave myocardial infarction, non-Q-wave myocardial infarction, death, need for bypass surgery, need for emergency bypass surgery,or need for repeat coronary angioplasty.